CLINICAL TRIAL: NCT01505231
Title: Vasopressin Versus Norepinephrine for the Management of Shock After Cardiac Surgery
Acronym: VaNCS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ludhmila Abrahão Hajjar, principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0352/08
Record Dates: First submitted 2012-01-02; First posted 2012-01-06 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Shock
Keywords: Shock; norepinephrine; vasopressin; cardiac surgery
MeSH Terms: conditions — Shock; Diabetes Insipidus | interventions — Vasopressins; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Norepinephrine group (Active Comparator): Blinded norepinephrine
  Interventions: Drug: Norepinephrine
- Vasopressin Group (Active Comparator): Blinded vasopressin
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Vasopressin — Blinded Vasopressin will be started if there is persistent hypotension, characterized by mean arterial pressure <65 mmHg after fluid replacement.
  Arms: Vasopressin Group
Drug: Norepinephrine — Blinded Norepinephrine will be started if there is persistent hypotension, characterized by mean arterial pressure <65 mmHg after fluid replacement
  Arms: Norepinephrine group

SUMMARY:
Vasoplegic syndrome after cardiac surgery is a common complication after cardiac surgery, with negative impact on patient outcomes and hospital costs. Pathogenesis of vasodilatory phenomenon after cardiac surgery remains a matter of controversy. Loss of vascular tone can be partly explained by the depletion of neurohypophyseal arginine vasopressin stores. The investigators hypothesized that the use of arginine vasopressin would be more effective on treatment of shock after cardiac surgery than norepinephrine, decreasing the composite end point of mortality and severe morbidity.

ELIGIBILITY:
Inclusion Criteria:

* need vasopressor support

Exclusion Criteria:

* younger than 18 years;
* surgery without cardiopulmonary bypass;
* emergency procedure;
* ascending and descending thoracic aortic procedures;
* left ventricular aneurysm resection; enrollment in another study;
* pregnancy;
* neoplasm;
* Raynaud's phenomenon, systemic sclerosis or vasospastic diathesis;
* severe hyponatremia (Na<130mEq/L);
* acute mesenteric ischemia;
* acute myocardial infarction;
* cardiogenic shock; and refusal to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-02 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of major morbidity according to Society of Thoracic Surgery | 30 days
  The primary end point is major morbidity according to STS (30-days mortality, mechanical ventilation > 48 hours, mediastinitis, surgical reexploration, stroke, acute renal failure)

SECONDARY OUTCOMES:
Hemodynamic effects | 28 days
  the time to attainment of hemodynamic stability ; the changes in hemodynamic variables; and the use of dobutamine or other inotropic agents.
occurence of adverse events and safety | 28 days
  Adverse events were categorized as arrhythmias, myocardial necrosis, skin necrosis, ischemia in limbs or distal extremities, or secondary infections
Time on mechanical ventilation | 30 days
  Days on mechanical ventilation during 30-days after surgery.
Incidence of infecction | 30-days
  Incidence of new infecction, sepsis, severe sepsis or septic shock in 30 days after surgery.
Length of ICU and Hospital stay | 90 days
  Compare between groups the period of time (days) that patients were in ICU and in Hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] O'Callaghan DJ, Gordon AC. What's new in vasopressin? Intensive Care Med. 2015 Dec;41(12):2177-9. doi: 10.1007/s00134-015-3849-3. Epub 2015 May 7. No abstract available. PMID 25947955